CLINICAL TRIAL: NCT03002142
Title: Auditory Rehabilitation With Hearing Aids and Cognition in Alzheimer Patients
Brief Title: Auditory Rehabilitation and Cognition in Alzheimer Patients
Acronym: RACO-MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRI15-DB/RACO-MA
Record Dates: First submitted 2016-03-16; First posted 2016-12-23 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer's Disease; Hearing Loss
Keywords: Alzheimer; Hearing loss; Cognition; Quality of life; Hearing aids
MeSH Terms: conditions — Alzheimer Disease; Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with hearing aids (Experimental): Patients fitted with functional hearing aids (Phonak Audéo BR)
  Interventions: Device: Hearing aids
- Patients treated with placebo device (Placebo Comparator): Patients fitted with non-functional hearing aids
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Hearing aids — Phonak Audéo B-R (Target V 5.0)
  Arms: Patients treated with hearing aids
Device: Placebo — Phonak Audéo B-R (Target V 5.0) without amplification
  Other Names: Non functional hearing aids
  Arms: Patients treated with placebo device

SUMMARY:
Alzheimer disease is a neurodegenerative disease. Recent studies suggest that subjects with hearing loss are more likely to develop Alzheimer's disease. Hearing loss can be consecutive to presbycusis and/or to central auditory dysfunction.

Standard audiometric measures with pure tone and speech intelligibility allow the diagnosis of presbycusis. However, to demonstrate central auditory dysfunction, specific audiometric tests as noisy and/or dichotic tests, are needed.

Actually, no consensus exists to investigate hearing loss in people with Alzheimer's disease; therefore hearing loss may be an early manifestation of Alzheimer's disease. Until now, investigations and clinical procedure related to the diagnosis of Alzheimer's disease ignored the hearing ability of the patient. However, the major part of care management and investigations implies the patient's communication ability with caregivers. Hearing loss may be one of the most unrecognized deficit in subjects with Alzheimer's disease. Auditory rehabilitation with hearing aids could benefit to the patient to decrease cognitive decline but this management must be investigate during longitudinal studies in order to demonstrate their efficiency and need to be compared with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer patient
* Mini Mental state examination= 15-25 or mild cognitive impairment
* Over 65 yo
* Sensorineural hearing loss with pure tone average over 30 dB
* Language: French
* Able to sign the consent
* Affiliated to the French social security

Exclusion Criteria:

* Conductive hearing loss
* Retrocochlear hearing loss
* History of neurological disorders with consequences in hearing loss (vascular accident; brain surgery, cerebral tumors, head trauma with loss consciousness)
* patient included in another study
* French no spoken
* chronic used of drugs or alcohol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
Changing score in Cognitive functions measured with Alzheimer's Disease Assessment Scale-cognitive scale | Change before and one year after the fitting with device
  French scale validated by the french society of geriatry

SECONDARY OUTCOMES:
air and bone auditory thresholds (dB HL) measured at 500, 1000, 2000, 3000 and 4000 Hz | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  Tonal audiometry
Speech recognition threshold (dB HL) measured by speech audiometry | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  Speech audiometry
Speech Discrimination Test (%) measured by speech audiometry | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  Speech audiometry
Dichotic test measured with audiometry | From 1 to 90 days prior the fitting with device
  Speech audiometry
Amplification with hearing aids or placebo devices measured by tonal and speech audiometry (dB HL) | 6 months after the fitting with device, 12 months after the fitting with device
  Audiometry
Devices tolerance measured with number of hours per day with hearing aids | 6 months after the fitting with device, 12 months after the fitting with device
  Audiometry
Objective auditory thresholds measured with auditory brainstem responses (ms) | 6 months after the fitting with device, 12 months after the fitting with device
  in case of uncooperative patients or to confirm tonal audiometry
Objective auditory thresholds measured by Auditory steady state responses (in dB eHL) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  in case of uncooperative patients or to confirm tonal audiometry
Mini Mental State Examination (30 items, total score from 0-30) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Hearing Handicap Inventory for Elderly measured by questionnaire (10 items, total score from 0-40) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Hearing loss impact scale in adults measured by 2 questionnaire (Abbreviated Profile of Hearing Aid Benefit, 24 items) and Impact of hearing loss in adults (20 items, total score from 0-200) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Quality of life-Alzheimer disease scale measured by questionnaire (total score from 13-52) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Assessing caregiver burden measured by Zarit scale (22 items, total score from 0-88) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Depression in the elderly measured by Geriatric depression scale (30 items, total score from 0-30) | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Executive functions measured by trail making test | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Working memory and processing speed measured by Wechsler Adult Intelligence Scale | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Speech comprehension measured by Beauregard tests | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version
Hearing aids tolerance measured by Glagow hearing-aid benefit questionnaire | From 1 to 90 days prior the fitting with device, 6 months after the fitting with device, 12 months after the fitting with device
  French validated version

CONTACTS AND LOCATIONS:
Overall Officials: DAVID BAKHOS, MCU-PU, Principal Investigator — University Hospital, Tours
Locations (1):
- University Hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided